CLINICAL TRIAL: NCT03266562
Title: Assessment of the Heterogeneity of Estrogen Receptor Expression in Patients With Estrogen Receptor Positive Breast Cancer Using F-18 Fluoroestradiol and High Resolution Positron Emission Mammography
Brief Title: Estrogen Receptor Expression in Breast Cancer - Assessed With Positron Emission Mammography
Acronym: PEM-FES
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit patients due to competing studies
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael O'Connor, consultant on medical physics, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-007764
Record Dates: First submitted 2016-11-30; First posted 2017-08-30 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Breast Neoplasm
Keywords: Positron Emission Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- FES vs FDG (Other): All patients will undergo two PEM studies, one with F-18 FDG and the second with F-18 FES. Co-registration of the PEM images from F-18 FDG and F-18 FES will be used to assess the heterogeneity of uptake of the F-18 FES relative to that of F-18 FDG. Heterogeneity of ER expression in the tumor will be determined by immunohistochemistry on the pathologic tissue
  Interventions: Diagnostic Test: F-18 FES; Diagnostic Test: F-18 FDG

INTERVENTIONS:
Diagnostic Test: F-18 FES — Evaluate uptake of F-18 FES in breast tissue
Diagnostic Test: F-18 FDG — Evaluate uptake of F-18 FDG in breast tissue

SUMMARY:
The primary objective of this study is to determine the correlation between the distribution of F-18 FES within ER+ breast tumors as seen on Positron Emission Mammography (PEM) images of the breast, and the distribution of cells stained ER+ within the tumor by immunohistochemistry (IHC) measurements at surgical pathology. The secondary aim is to determine if the correlation (or lack of) between F-18 FES uptake and F-18 FDG uptake as imaged by PEM, is an accurate representation of the heterogeneity of ER expression in the tumor.

DETAILED DESCRIPTION:
This pilot study will recruit up to 20 patients with newly diagnosed ER+ breast cancer who have recently undergone or are scheduled to undergo a clinically-indicated breast MRI examination and are scheduled for surgical excision of the breast cancer. All patients will undergo two PEM studies, one with F-18 FDG and the second with F-18 FES. As F-18 FES is not an FDA-approved radiopharmaceutical, this FES study will be performed under an investigator IND cross-referenced to the National Cancer Institute IND 79,005 for F-18 FES. A time interval of 6-8 hours will be required between performance of the F-18 FDG study and the F-18 FES study. All patients will have the 2 PEM studies within 30 business days of the clinically indicated MRI. See Study Schema shown below. Subjects must meet the following eligibility criteria:

1. Postmenopausal women, as defined by a. Lack of menstrual periods for ≥ 12 months b. For women with prior hysterectomy and age < 60, a serum FSH level within the postmenopausal range
2. Histologic proof of invasive breast carcinoma that is ER positive per ASCO/CAP guidelines (staining in ≥ 1% of cells by immunohistochemistry)
3. Extent of disease confirmed, or to be confirmed, on a clinical contrast-enhanced breast MRI examination
4. Minimum size criteria for index cancer of 10 mm as measured on mammogram, ultrasound, or MRI.
5. Planned surgical excision of the breast cancer at Mayo Clinic, Rochester

Study participants will be consented prior to undergoing the PEM studies. The order in which the PEM and MRI studies are performed will NOT be randomized, and will be dictated by patient schedule. Co-registration of the PEM images from F-18 FDG and F-18 FES will be used to assess the heterogeneity of uptake of the F-18 FES relative to that of F-18 FDG. Heterogeneity of ER expression in the tumor will be determined by immunohistochemistry on the pathologic tissue and findings will then be correlated with the ratio of activity in the co-registered images of F-18 FES and F-18 FDG. An integrated interpretation of the MRI and PEM images will be performed to match lesions seen on the three scans and will be made available to the ordering physician and surgeon.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will be offered enrollment if the time interval between initial diagnosis and surgery allows for performance of the PEM studies with both F18 FDG and F-18 FES, and they meet the following criteria:

* Postmenopausal women, as defined by

  * Lack of menstrual periods for ≥ 12 months
  * For women with prior hysterectomy and age < 60, a serum FSH level within the postmenopausal range
* Histologic proof of invasive breast carcinoma that is ER positive per ASCO/CAP guidelines (staining in ≥ 1% of cells by immunohistochemistry)
* Extent of disease confirmed, or to be confirmed, on a clinical contrast-enhanced breast MRI examination
* Minimum size criteria for index cancer of 10 mm as measured on mammogram, ultrasound, or MRI.
* Planned surgical excision of the breast cancer at Mayo Clinic, Rochester

Exclusion Criteria:

Patients are excluded if they meet any of the following criteria:

* Premenopausal
* Unable to undergo PEM scanning (weight limit of 300 lbs. on PEM system or inability to lie prone for 30 minutes)
* Total serum bilirubin > 1.5 x upper limit of normal (abnormal hepatic metabolism may interfere with FES hepatic excretion),
* Serum creatinine > 1.5 x upper limit of normal
* Patients who have received, are currently receiving, or planning to receive neoadjuvant systemic therapy prior to surgical excision
* Patients who will undergo core needle biopsy of the breast or axilla between the breast MRI and investigational PEM studies. NOTE: Axillary ultrasound with or without fine needle aspiration of an axillary mass or lymph node is allowed.
* Patients with breast implants?

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
correlation of FES and estrogen receptors | 1 year
  The primary objective of this study is to determine the correlation between F-18 FES uptake on PEM, and distribution of ER+ tissue on pathology

SECONDARY OUTCOMES:
correlation of FES and FDG in breast tumors | 1 year
  The secondary aim is to determine if the correlation (or lack of) between F-18 FES uptake and F-18 FDG uptake as imaged by PEM, is an accurate representation of the heterogeneity of ER expression in the tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Michael K O'Connor, Ph.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials